CLINICAL TRIAL: NCT05849909
Title: Evaluation of the Vulnerable Carotid Atherosclerotic Plaque: A Clinical Multicenter Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: huang pintong (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor-Investigator, huang pintong, Director of Ultrasound Department, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Other Study IDs: 2023-0402
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Ultrasound

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stable Carotid Atherosclerotic Plaques
- Unstable Carotid Atherosclerotic Plaques

SUMMARY:
Evaluation of carotid plaque vulnerability based on ultrasound imaging features， proteomics and metabolomics: a clinical multicenter study

DETAILED DESCRIPTION:
Carotid artery plaque tissue specimen for proteomics. Blood were collect for metabolomics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the CEA surgical indications;
2. Age>18 years old;
3. Patients who sign informed consent forms

Exclusion Criteria:

1. Those with severe calcification of plaques and obvious acoustic shadows, and poor image quality;
2. Contraindications to ultrasound contrast, such as those who are allergic to contrast agents;
3. Intracardiac right to left shunt;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing carotid endarterectomy
Sampling Method: Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2024-04-18 (Estimated)

PRIMARY OUTCOMES:
ultrasound | 2023.05
  B mode

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ultrasound, Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided